CLINICAL TRIAL: NCT07027098
Title: Retinal Displacement After Pars Plana Vitrectomy for Macula Involving Retinal Detachment: A Randomised Prospective Study Evaluating the Role of Intraoperative Perfluorocarbon Liquids
Brief Title: Pars Plana Vitrectomy and Influence of Perfluorocarbon Liquids on Retinal Displacement
Acronym: PAVILION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 327806 (129-06-23)
Record Dates: First submitted 2025-02-25; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-02

CONDITIONS: Retinal Displacement After Retinal Detachment Surgery
Keywords: Retinal displacement; retinal detachment; Heavy liquid; perfluorocarbon liquids
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Intervention Model Description: This trial is designed as a double-blind parallel arm randomised control trial. The trial is designed to show superiority regarding the use of PFCL intraoperatively as compared to without, when relevant to outcomes such as retinal displacement. It will be double blind because neither the participants nor the researchers assessing the outcomes will know what treatment each participant received; the surgeons providing treatment will unavoidably know this.
Who Masked: Participant
Masking Description: All participants will be masked to the surgical arm they are placed in, as will the investigators examining for retinal displacement (primary outcome).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinal Detachment Surgery (Vitrectomy) With Perflurocarbon liquid use. (Experimental): Standard retinal detachment surgery (vitrectomy) with the use of Perflurocarbon liquid (PFCL) to stabilise macular during surgery and drainage of subretinal fluid. PFCL is then fully removed before the end of surgery.
  Interventions: Procedure: Perflurocarbon liquid
- Retinal Detachment Surgery (Vitrectomy) Without Perflurocarbon liquid use. (Active Comparator): Standard retinal detachment surgery (vitrectomy) without the use of Perflurocarbon liquid (PFCL).
  Interventions: Procedure: Without Perflurocarbon liquid

INTERVENTIONS:
Procedure: Perflurocarbon liquid — Used to facilitate surgery of retinal detachment to stabilise macular during surgery.
  Arms: Retinal Detachment Surgery (Vitrectomy) With Perflurocarbon liquid use.
Procedure: Without Perflurocarbon liquid — Standard retinal detachment surgery (vitrectomy) without the use of Perflurocarbon liquid (PFCL).
  Arms: Retinal Detachment Surgery (Vitrectomy) Without Perflurocarbon liquid use.

SUMMARY:
Rhegmatogenous retinal detachment (RRD) is an acute, sight threatening condition, with an incidence of approximately 10 per 100,000 people. Surgical interventions for treating RRD include pars plana vitrectomy (PPV), which currently represents the main adopted surgical choice. Main outcomes of successful RRD surgery have mainly been represented by anatomical retinal reattachment and best-corrected visual acuity (BCVA). Despite successful surgery, patients with mac-off RRD often report postoperative visual complaints of distortion such as metamorphopsia and scotomas in their central visual field, with great variability.

Major advances in retinal imaging including wide-field optical coherence tomography (OCT) and fundus autofluorescence (FAF) allowed to investigate morphological changes after RRD surgery. The concept of retinal displacement - where the retina has reattached but the exact location has shifted, as evidenced by retinal vessel printing shown on post operative retinal imaging.

Postoperative retinal displacement has been observed to occur with different frequency in relationship to variables including postoperative tamponade, surgical technique, and intraoperative use of perfluorocarbon liquids (PFCL). The investigators hope to formally study the impact of intraoperative use of PFCL, which is used as an aid during surgery to help flatten and position the retina, on retinal displacement. This will help us better understand the impact of this tool on outcomes both objectively through retinal imaging, and subjectively through visual outcomes including visual acuity and measures of distortion and other visual disturbances.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment (RRD) is an acute, sight threatening condition, resulting from the separation of the neurosensory retina from the underlying retinal pigment epithelium (RPE). It is caused by at least one retinal break and recruitment of intraocular fluid into the subretinal space. Surgical interventions for treating RRD include pars plana vitrectomy (PPV), which currently represents the most widely adopted surgical choice, scleral buckling (SB) and pneumatic retinopexy (PnR).

Significant visual loss is the main complaint of patients with macula-involving RRD (MIRD). Hence, the main outcomes of successful RRD surgery have historically been represented by postoperative anatomical retinal reattachment and best-corrected visual acuity (BCVA). However, despite successful surgery, patients with MIRD often report postoperative visual complaints of distortion such as metamorphopsia, aniseikonia and scotomas in their central visual field, with great variability.

Major advances in retinal imaging contributed to provide a better understanding of postoperative visual complaints after surgery for RRD. In particular, optical coherence tomography (OCT) highlighted drop-out of the ellipsoid zone (EZ) or outer and inner retinal folds in the macula area. However, only more recently, hyperautofluorescent lines, also called Retinal Vessel Printing (RVP), adjacent to the retinal blood vessels, were noted on autofluorescence imaging in patients who underwent RRD surgery. This finding is believed to be secondary to unintentional retinal displacement after RRD surgery and may serve as a surrogate anatomical marker of postoperative metamorphopsia and central scotomas.

Postoperative retinal displacement is potentially influenced by several variables including intraocular tamponade, adopted surgical technique, intraoperative use of perfluorocarbon liquids (PFCL) and postoperative posture. The effect of PFCL on retinal displacement is currently unknown due to lack of RCTs and significant limitations of previous research. Therefore, the aim of this RCT is to investigate the role of intraoperative PFCL on postoperative retinal displacement in patients with MIRD undergoing PPV with immediate postoperative face-down posture.

The investigators aim to evaluate whether intraoperative PFCL affects the incidence and patterns of postoperative retinal displacement. As secondary outcomes, this RCT will also investigate the effect of intraoperative use of PFCL on functional outcomes, e.g. BCVA, metamorphopsia and aniseikonia. All patients participating in the trial will be randomly allocated to having surgery either with or without the use of PFCL, and will be followed up regularly after surgery for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, or older.
* Diagnosis of primary MIRD with posterior vitreous detachment, and fovea off (confirmed with OCT)
* Surgeons' decision that the patient is eligible for using gas as postoperative tamponade.
* The surgeon is confident to proceed with surgery with or without the use of intraoperative PFCL

Exclusion Criteria:

* Previous RRD and/or RRD surgery in the study eye
* Decision to use adjunct scleral buckle
* Decision to use silicone oil as tamponade
* Retinal detachment with macula on
* Patients with other retinal pathologies causing permanent structural changes to the retina in the study eye, such as diabetic retinopathy (assessed above background, or any diabetic maculopathy), previous vascular occlusion (artery or vein occlusion), macula dystrophy, among others
* Previous vitreoretinal surgery in the study eye
* Inability to come for follow ups up to 3 months
* Inability to take FAF and OCT imaging due to neck stiffness or other medical issue
* Mental incapacity
* Patient is unwilling or unable to follow or comply with all study related procedures or to sign informed consent form.
* Contraindications for PFCL
* Previous enrollment in a clinical trial involving retinal diseases and/or treatments
* Media opacity leading to poor quality retinal images (not including post operative significant cataract. See section 7.11)
* Patient inability to posture following surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Retinal Displacement | 3 months post operation
  Number of patients with presence of retinal displacement on post operative retinal imaging (FAF) between groups with PFCL use and without PFCL use.

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity | Baseline, 2 weeks, 3 months, and 6 months (at discretion of research team, see protocol)
  Average change in visual acuity (BCVA) in groups with PFCL and without PFCL use
Aniseikonia | 3 months post operation
  Average Awaya Test score comparison between groups with PFCL and without PFCL use.
Metamorphopsia | 3 months post operation
  Average M-CHARTS score comparison between groups with PFCL use and without PFCL use.
Quantification of retinal displacement | 3 months post operation
  Retinal displacement distance as measured on retinal imaging (FAF) in millimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sabatino, Principal Investigator — Norwich University Hospitals NHS Foundation Trust,
Locations (1):
- Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom